CLINICAL TRIAL: NCT04209114
Title: A Phase 3, Randomized, Study of Neoadjuvant and Adjuvant Nivolumab Plus Bempegaldesleukin (NKTR-214), Versus Nivolumab Alone Versus Standard of Care in Participants With Muscle-Invasive Bladder Cancer (MIBC) Who Are Cisplatin Ineligible
Brief Title: A Study of Nivolumab Plus Bempegaldesleukin (Bempeg/NKTR-214) vs Nivolumab Alone vs Standard of Care in Participants With Bladder Cancer That May Have Invaded The Muscle Wall of the Bladder and Who Cannot Get Cisplatin, A Type of Medicine Given To Treat Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA045-009; 2018-002676-40 (EudraCT Number); 18-214-13 (Other: Nektar Therapeutics)
Record Dates: First submitted 2019-12-20; First posted 2019-12-23 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Bladder Cancer; Bladder Tumor; Muscle-Invasive Bladder Cancer
Keywords: immunotherapy; NKTR-214; nivolumab; bempeg
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Nivolumab; Cystectomy; bempegaldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Combination Therapy (Experimental): Neoadjuvant (pre-surgical treatment) nivolumab + bempeg, followed by radical cystectomy (RC), followed by adjuvant (post-surgical treatment) nivolumab + bempeg
  Interventions: Biological: Nivolumab; Procedure: Radical cystectomy (RC); Biological: Bempegaldesleukin
- Arm B: Monotherapy (Experimental): Neoadjuvant nivolumab, followed by RC, followed by adjuvant nivolumab
  Interventions: Biological: Nivolumab; Procedure: Radical cystectomy (RC)
- Arm C: Standard-of-care (Other): RC alone, without neoadjuvant or adjuvant therapy
  Interventions: Procedure: Radical cystectomy (RC)

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Arm A: Combination Therapy; Arm B: Monotherapy
Procedure: Radical cystectomy (RC) — Surgical removal of the bladder
Biological: Bempegaldesleukin — Specified dose on specified days
  Other Names: BMS-986321; NKTR-214; Bempeg
  Arms: Arm A: Combination Therapy

SUMMARY:
The purpose of the study is to see if treatment with nivolumab plus bempegaldesleukin or nivolumab alone, before and after surgery to remove the bladder, is more effective than surgery alone in participants with high-risk urothelial cancer, including muscle-invasive bladder cancer who are not able to receive cisplatin chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Urothelial carcinoma (UC) of the bladder, clinical stage T2-T4aN0, M0 or T1-T4aN1, M0, diagnosed at transurethral resection of bladder tumor (TURBT)
* Must be deemed eligible for Radical Cystectomy (RC) by urologist, and must agree to undergo RC. For arms A and B, participants must agree to undergo RC after completion of neoadjuvant therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Cisplatin-ineligible participants will be defined by any one of the following criteria:

  i) Impaired renal function (glomerular filtration rate [GFR] ≥ 30 but < 60 mL/min) ii) GFR should be assessed by direct measurement (ie, creatinine clearance) or, if not available, by calculation from serum/plasma creatinine (Cockcroft-Gault formula) iii) Common Terminology Criteria for Adverse Events (CTCAE) version 5, ≥ Grade 2 hearing loss (assessed per local SOC).

iv) CTCAE version 5, ≥ Grade 2 peripheral neuropathy.

* Documented Left Ventricular Ejection Fraction (LVEF) more than 45%

Exclusion Criteria:

* Clinical evidence of ≥ N2 or metastatic bladder cancer
* Prior systemic therapy, radiation therapy, or surgery for bladder cancer other than TURBT or biopsies is not permitted. Prior Bacillus Calmette-Guerin (BCG) or other intravesicular treatment of non-muscle invasive bladder cancer (NMIBC) is permitted if completed at least 6 weeks prior to initiating study treatment.
* Evidence of urothelial carcinoma (UC) in upper urinary tracts (ureters or renal pelvis) or history of previous MIBC
* History of pulmonary embolism (PE), deep vein thrombosis (DVT), or prior clinically significant venous or non-CVA(cerebrovascular accident)/TIA (Transient ischemic attack) arterial thromboembolic event
* Known cardiovascular history, including unstable or deteriorating cardiac disease within the previous 12 months (including unstable angina or myocardial infarction, congestive heart failure or uncontrolled clinically significant arrhythmias)

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (116):
- United States (15):
  - Local Institution - 0080, Gilbert, Arizona
  - Local Institution - 0136, Tucson, Arizona
  - Local Institution - 0029, La Jolla, California
  - Local Institution - 0015, Orange, California
  - Local Institution - 0002, Iowa City, Iowa
  - Local Institution, Rochester, Minnesota
  - Local Institution - 0006, New Brunswick, New Jersey
  - Local Institution - 0004, Buffalo, New York
  - Local Institution - 0009, The Bronx, New York
  - Local Institution - 0005, Allentown, Pennsylvania
  - Local Institution - 0007, Charleston, South Carolina
  - Local Institution - 0139, Houston, Texas
  - Local Institution - 0023, Temple, Texas
  - Local Institution - 0122, Gig Harbor, Washington
  - Local Institution - 0102, Seattle, Washington
- Argentina (6):
  - Local Institution - 0096, Capital Federal, Buenos Aires
  - Local Institution - 0028, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0124, La Plata, Buenos Aires
  - Local Institution - 0027, Capital Federal, Distrito Federal
  - Local Institution - 0174, Rosario, Santa Fe Province
  - Local Institution - 0097, Córdoba
- Australia (5):
  - Local Institution - 0137, Gosford, New South Wales
  - Local Institution - 0158, Ballarat, Victoria
  - Local Institution - 0157, Fitzroy, Victoria
  - Local Institution - 0011, Heidelberg, Victoria
  - Local Institution - 0013, Murdoch, Western Australia
- Austria (3):
  - Local Institution - 0148, Graz
  - Local Institution - 0123, Vienna
  - Local Institution - 0150, Vienna
- Belgium (5):
  - Local Institution - 0083, Wilrijk, Antwerpen
  - Local Institution - 0101, Brussels, Brussels Capital
  - Local Institution - 0098, Edegem
  - Local Institution - 0068, Ghent
  - Local Institution - 0100, Liège
- Brazil (7):
  - Local Institution - 0177, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0039, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0176, Barretos, São Paulo
  - Local Institution - 0037, Jaú, São Paulo
  - Local Institution - 0038, São Paulo, São Paulo
  - Local Institution - 0041, Rio de Janeiro
  - Local Institution - 0040, São Paulo
- Canada (3):
  - Local Institution - 0082, Oshawa, Ontario
  - Local Institution - 0018, Québec, Quebec
  - Local Institution - 0036, Sherbrooke, Quebec
- China (7):
  - Local Institution - 0204, Chongqing, Chongqing Municipality
  - Local Institution, Xiamen, Fujian
  - Local Institution, Zhengzhou, Henan
  - Local Institution, Wuhan, Hubei
  - Local Institution, Changsha, Hunan
  - Local Institution, Taiyuan, Shan1xi
  - Local Institution, Jinan, Shandong
- Czechia (3):
  - Local Institution - 0022, Olomouc
  - Local Institution - 0021, Prague
  - Local Institution - 0020, Prague
- France (15):
  - Local Institution - 0077, Avignon
  - Local Institution - 0091, Bordeaux
  - Local Institution - 0151, Clermont-Ferrand
  - Local Institution - 0059, La Roche-sur-Yon
  - Local Institution - 0071, Lyon
  - Local Institution - 0057, Marseille
  - Local Institution - 0075, Montpellier
  - Local Institution - 0070, Nice
  - Local Institution - 0062, Paris
  - Local Institution - 0060, Paris
  - Local Institution - 0064, Quimper
  - Local Institution - 0161, Reims
  - Local Institution - 0058, Strasbourg
  - Local Institution - 0056, Suresnes
  - Local Institution - 0074, Tours
- Germany (12):
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Local Institution - 0117, Düsseldorf
  - Local Institution - 0119, Erlangen
  - Local Institution - 0050, Essen
  - Local Institution - 0052, Hamburg
  - Local Institution - 0051, Hamburg
  - Local Institution - 0049, Herne
  - Local Institution - 0045, Jena
  - Local Institution - 0053, Lübeck
  - Local Institution - 0113, Münster
  - Local Institution - 0048, Nuremberg
  - Local Institution - 0046, Tübingen
- Greece (4):
  - Local Institution - 0178, Athens
  - Local Institution - 0088, Athens
  - Local Institution - 0033, Chaïdári
  - Local Institution - 0035, Thessaloniki
- Israel (3):
  - Local Institution - 0129, Haifa
  - Local Institution - 0131, Tel Aviv
  - Local Institution - 0130, Tel Litwinsky
- Italy (7):
  - Local Institution - 0149, Florence
  - Local Institution - 0162, Milan
  - Local Institution - 0025, Milan
  - Local Institution, Pavia
  - Local Institution - 0026, Pisa
  - Local Institution - 0065, Roma
  - Local Institution - 0044, Rozzano
- Mexico (4):
  - Local Institution - 0154, La Paz, BAJA Californa SUR
  - Local Institution - 0132, Mexico City, Mexico City
  - Local Institution - 0160, Mexico City, Mexico City
  - Local Institution - 0133, Monterrey, Nuevo León
- Local Institution - 0069, Amsterdam, Netherlands
- Poland (2):
  - Local Institution - 0167, Biała Podlaska
  - Local Institution - 0054, Warsaw
- Russia (2):
  - Local Institution, Omsk
  - Local Institution, Saint Petersburg
- Spain (9):
  - Local Institution - 0104, A Coruña
  - Local Institution - 0106, Badalona
  - Local Institution - 0110, Barcelona
  - Local Institution - 0109, Córdoba
  - Local Institution - 0105, Madrid
  - Local Institution - 0108, Madrid
  - Local Institution - 0103, Madrid
  - Local Institution - 0107, Santander
  - Local Institution - 0111, Seville
- United Kingdom (3):
  - Local Institution, Stevenage, Hertfordshire
  - Local Institution - 0085, Leicester
  - Local Institution - 0042, London

IPD SHARING:
Plan to Share IPD: Yes
Individual patient level data from this study may be shared with qualified researchers, upon request, following the timelines and process detailed on https://www.bms.com/researchers-and-partners/independent-research/data-sharing-request-process.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/home

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per Protocol Amendment 04, participants who are currently receiving bempegaldesleukin plus nivolumab in Arm A are required to discontinue bempegaldesleukin and may continue to receive nivolumab monotherapy.
Groups:
- Arm A: Nivolumab + Bempegaldesleukin: Bempegaldesleukin 0.006 mg/kg once every 3 weeks plus nivolumab 360 mg once every 3 weeks for 3 cycles as neoadjuvant therapy, followed by Radical Cystectomy, followed by bempegaldesleukin 0.006 mg/kg once every 3 weeks plus nivolumab 360 mg once every 3 weeks up to an additional 12 cycles.
- Arm B: Nivolumab: Nivolumab 360 mg once every 3 weeks for 3 cycles as neoadjuvant therapy, followed by Radical Cystectomy, followed by nivolumab 360 mg once every 3 weeks up to an additional 12 cycles.
- Arm C: Standard of Care: Standard of care therapy, with cystectomy alone, without neoadjuvant or adjuvant therapy.
Period: Pre-Treatment Phase
Arm/Group | Arm A: Nivolumab + Bempegaldesleukin | Arm B: Nivolumab | Arm C: Standard of Care
Started (Randomized) | 37 | 37 | 40
Completed (Treated) | 37 | 37 | 32
Not Completed | 0 | 0 | 8
Not completed — Completed without radical cystectomy | 0 | 0 | 5
Not completed — Other reasons | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Participant withdrew consent | 0 | 0 | 1
Period: Treatment Phase
Arm/Group | Arm A: Nivolumab + Bempegaldesleukin | Arm B: Nivolumab | Arm C: Standard of Care
Started (Treated) | 37 | 37 | 32
Completed | 15 | 13 | 32
Not Completed | 22 | 24 | 0
Not completed — Other reasons | 5 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Participant withdrew consent | 1 | 0 | 0
Not completed — Adverse event unrelated to study drug | 1 | 5 | 0
Not completed — Death | 4 | 1 | 0
Not completed — Study drug toxicity | 4 | 6 | 0
Not completed — Disease progression | 6 | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Nivolumab + Bempegaldesleukin | Arm B: Nivolumab | Arm C: Standard of Care | Total
Number analyzed (Participants) | 37 | 37 | 40 | 114
Age, Continuous [Median (Standard Deviation); unit: Years] | 73.0 (8.8) | 72.0 (7.5) | 74.5 (8.4) | 74.0 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 9 | 22
  Male | 31 | 30 | 31 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 36 | 35 | 36 | 107
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) Rate- Nivolumab + Bempegaldesleukin Compared to Standard of Care
Description: Pathologic Complete Response (pCR) is defined as the percentage of randomized participants with absence of any cancer in pathology specimens after radical cystectomy, based on blinded independent pathology review (BIPR). Participants who do not undertake surgery will be counted as non-pCR.
Time Frame: From time of radical cystectomy up to 100 days after last treatment (up to approximately 17 months)
Population: All randomized participants in Arms A and C
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Nivolumab + Bempegaldesleukin | Arm C: Standard of Care
Number analyzed (Participants) | 37 | 40
Percentage of participants | 10.8 [3.0 to 25.4] | 2.5 [0.1 to 13.2]

2. Primary Outcome: Event Free Survival (EFS) - Nivolumab + Bempegaldesleukin Compared to Standard of Care
Description: Event Free Survival (EFS) is defined as the time from randomization to any of the following events: progression of disease that precludes surgery, local or distant recurrence based on blinded independent committee review (BICR) assessments, or death due to any cause.
  Participants who did not have an EFS event will be censored on the date of their last evaluable tumor assessment (imaging or biopsy) or at the date of radical surgery whichever occur last. Participants who did not have any baseline tumor assessments (imaging or biopsy) and did not undergo radical cystectomy for other reason than worsening/progression of disease will be censored on their date of randomization. Participants who did not have any on study tumor assessments (imaging or biopsy) and did not die will be censored on their date of radical cystectomy (or randomization date if no radical cystectomy performed).
Time Frame: From randomization up to first EFS event (up to approximately 30 months)
Population: All randomized participants in Arms A and C
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivolumab + Bempegaldesleukin | Arm C: Standard of Care
Number analyzed (Participants) | 37 | 40
Months | 22.11 [8.21 to NA] — Upper limit not calculated due to insufficient number of events. | 15.18 [11.63 to NA] — Upper limit not calculated due to insufficient number of events.

3. Secondary Outcome: Pathologic Complete Response (pCR) Rate - Nivolumab Compared to Standard of Care
Description: as for outcome 1
Time Frame: From time of radical cystectomy up to 100 days after last treatment (up to approximately 17 months)
Population: All randomized participants in Arms B and C
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm B: Nivolumab | Arm C: Standard of Care
Number analyzed (Participants) | 37 | 40
Percentage of participants | 10.8 [3.0 to 25.4] | 2.5 [0.1 to 13.2]

4. Secondary Outcome: Event Free Survival (EFS) - Nivolumab Compared to Standard of Care
Description: as for outcome 2
Time Frame: From randomization up to first EFS event (up to approximately 30 months)
Population: All randomized participants in Arms B and C
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B: Nivolumab | Arm C: Standard of Care
Number analyzed (Participants) | 37 | 40
Months | NA [10.84 to NA] — Median and upper limit not calculated due to insufficient number of events. | 15.18 [11.63 to NA] — Upper limit not calculated due to insufficient number of events.

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time between the date of randomization and the date of death. For those without documentation of death, OS will be censored on the last date the participant was known to be alive.
  OS was not calculated for Arm A and Arm B because the number of events did not meet the threshold due to early study termination. In lieu of OS, time to death is reported as a Post-Hoc endpoint.
Time Frame: From randomization to study completion, up to approximately 40 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivolumab + Bempegaldesleukin | Arm B: Nivolumab | Arm C: Standard of Care
Number analyzed (Participants) | 37 | 37 | 40
Months | NA [NA to NA] — Median, lower and upper limit not calculated due to insufficient number of events. | NA [NA to NA] — Median, lower and upper limit not calculated due to insufficient number of events. | 23.23 [14.36 to NA] — Upper limit not calculated due to insufficient number of events.

6. Post Hoc Outcome: Time to Death
Description: The amount of time in months from when participants were randomized until death. Survival was reported as time to death instead of overall survival by Kaplan-Meier analysis due to the small number of events at the time of early study completion.
Time Frame: From randomization to study completion, up to approximately 40 months
Population: All randomized participants
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A: Nivolumab + Bempegaldesleukin | Arm B: Nivolumab | Arm C: Standard of Care
Number analyzed (Participants) | 37 | 37 | 40
Months | 6.77 [3.2 to 18.4] | 9.43 [1.8 to 20.1] | 8.49 [1.6 to 23.2]

7. Secondary Outcome: The Number of Participants Experiencing Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: from first dose to 100 days following last dose (up to approximately 20 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab + Bempegaldesleukin | Arm B: Nivolumab | Arm C: Standard of Care
Number analyzed (Participants) | 37 | 37 | 32
Participants | 34 | 36 | 19

8. Secondary Outcome: The Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: from first dose to 100 days following last dose (up to approximately 20 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab + Bempegaldesleukin | Arm B: Nivolumab | Arm C: Standard of Care
Number analyzed (Participants) | 37 | 37 | 32
Participants | 15 | 18 | 14

9. Secondary Outcome: The Number of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation
Description: as for outcome 7
Time Frame: from first dose to 100 days following last dose (up to approximately 20 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab + Bempegaldesleukin | Arm B: Nivolumab | Arm C: Standard of Care
Number analyzed (Participants) | 37 | 37 | 32
Participants | 8 | 8 | 0

10. Secondary Outcome: The Number of Participants Experiencing Immune-Mediated Adverse Events (IMAEs)
Description: IMAEs are specific AEs that include pneumonitis, diarrhea/colitis, hepatitis, nephritis/renal dysfunction, rash, endocrine (adrenal insufficiency, hypothyroidism/thyroiditis, hyperthyroidism, diabetes mellitus, and hypophysitis), and other specific events, considered as potential immune-mediated events by investigator that meet the definition summarized below:
  * those occurring within 100 days of the last dose,
  * regardless of causality,
  * treated with immune-modulating medication (of note, endocrine AEs such as adrenal insufficiency, hypothyroidism/thyroiditis, hyperthyroidism, diabetes mellitus, and hypophysitis are considered IMAEs regardless of immune-modulating medication use, since endocrine drug reactions are often managed without immune-modulating medication).
  * with no clear alternate etiology based on investigator assessment, or with an immune-mediated component.
Time Frame: from first dose to 100 days following last dose (up to approximately 20 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab + Bempegaldesleukin | Arm B: Nivolumab | Arm C: Standard of Care
Number analyzed (Participants) | 37 | 37 | 32
Participants | 10 | 10 | 0

11. Secondary Outcome: Worst Grade Clinical Laboratory Values
Description: Clinical laboratory values by worst CTC grade are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose to 100 days following last dose (up to approximately 20 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab + Bempegaldesleukin | Arm B: Nivolumab | Arm C: Standard of Care
Number analyzed (Participants) | 37 | 37 | 32
Participants
  Hemoglobin: Grade 0 | 5 | 5 | 0
  Hemoglobin: Grade 1 | 23 | 23 | 2
  Hemoglobin: Grade 2 | 7 | 8 | 3
  Hemoglobin: Grade 3 | 1 | 1 | 1
  Hemoglobin: Grade 4 | 0 | 0 | 0
  Hemoglobin: Not Reported | 1 | 0 | 26
  Platelet Count: Grade 0 | 35 | 34 | 5
  Platelet Count: Grade 1 | 1 | 3 | 1
  Platelet Count: Grade 2 | 0 | 0 | 0
  Platelet Count: Grade 3 | 0 | 0 | 0
  Platelet Count: Grade 4 | 0 | 0 | 0
  Platelet Count: Not Reported | 1 | 0 | 26
  Leukocytes, Local Lab: Grade 0 | 33 | 35 | 6
  Leukocytes, Local Lab: Grade 1 | 2 | 2 | 0
  Leukocytes, Local Lab: Grade 2 | 0 | 0 | 0
  Leukocytes, Local Lab: Grade 3 | 1 | 0 | 0
  Leukocytes, Local Lab: Grade 4 | 0 | 0 | 0
  Leukocytes, Local Lab: Not Reported | 1 | 0 | 26
  Lymphocytes (Absolute), Local Lab: Grade 0 | 23 | 12 | 0
  Lymphocytes (Absolute), Local Lab: Grade 1 | 4 | 6 | 0
  Lymphocytes (Absolute), Local Lab: Grade 2 | 0 | 6 | 0
  Lymphocytes (Absolute), Local Lab: Grade 3 | 3 | 2 | 0
  Lymphocytes (Absolute), Local Lab: Grade 4 | 0 | 0 | 0
  Lymphocytes (Absolute), Local Lab: Not Reported | 7 | 11 | 32
  Absolute Neutrophil Count: Grade 0 | 31 | 36 | 0
  Absolute Neutrophil Count: Grade 1 | 4 | 1 | 0
  Absolute Neutrophil Count: Grade 2 | 0 | 0 | 0
  Absolute Neutrophil Count: Grade 3 | 0 | 0 | 0
  Absolute Neutrophil Count: Grade 4 | 1 | 0 | 0
  Absolute Neutrophil Count: Not Reported | 1 | 0 | 32
  Alkaline Phosphate, Local Lab: Grade 0 | 24 | 30 | 2
  Alkaline Phosphate, Local Lab: Grade 1 | 10 | 7 | 0
  Alkaline Phosphate, Local Lab: Grade 2 | 2 | 0 | 0
  Alkaline Phosphate, Local Lab: Grade 3 | 0 | 0 | 0
  Alkaline Phosphate, Local Lab: Grade 4 | 0 | 0 | 0
  Alkaline Phosphate, Local Lab: Not Reported | 1 | 0 | 30
  Aspartate Aminotransferase, Local Lab: Grade 0 | 31 | 30 | 2
  Aspartate Aminotransferase, Local Lab: Grade 1 | 5 | 6 | 0
  Aspartate Aminotransferase, Local Lab: Grade 2 | 0 | 1 | 0
  Aspartate Aminotransferase, Local Lab: Grade 3 | 0 | 0 | 0
  Aspartate Aminotransferase, Local Lab: Grade 4 | 0 | 0 | 0
  Aspartate Aminotransferase, Local Lab: Not Reported | 1 | 0 | 30
  Alanine Aminotransferase, Local Lab: Grade 0 | 26 | 30 | 2
  Alanine Aminotransferase, Local Lab: Grade 1 | 10 | 7 | 0
  Alanine Aminotransferase, Local Lab: Grade 2 | 0 | 0 | 0
  Alanine Aminotransferase, Local Lab: Grade 3 | 0 | 0 | 0
  Alanine Aminotransferase, Local Lab: Grade 4 | 0 | 0 | 0
  Alanine Aminotransferase, Local Lab: Not Reported | 1 | 0 | 30
  Total Bilirubin, Local Lab: Grade 0 | 33 | 35 | 2
  Total Bilirubin, Local Lab: Grade 1 | 2 | 2 | 0
  Total Bilirubin, Local Lab: Grade 2 | 1 | 0 | 0
  Total Bilirubin, Local Lab: Grade 3 | 0 | 0 | 0
  Total Bilirubin, Local Lab: Grade 4 | 0 | 0 | 0
  Total Bilirubin, Local Lab: Not Reported | 1 | 0 | 30
  Creatinine, Local Lab: Grade 0 | 11 | 13 | 5
  Creatinine, Local Lab: Grade 1 | 10 | 14 | 1
  Creatinine, Local Lab: Grade 2 | 12 | 9 | 0
  Creatinine, Local Lab: Grade 3 | 3 | 1 | 0
  Creatinine, Local Lab: Grade 4 | 0 | 0 | 0
  Creatinine, Local Lab: Not Reported | 1 | 0 | 26
  Hypernatremia: Grade 0 | 34 | 36 | 6
  Hypernatremia: Grade 1 | 2 | 1 | 0
  Hypernatremia: Grade 2 | 0 | 0 | 0
  Hypernatremia: Grade 3 | 0 | 0 | 0
  Hypernatremia: Grade 4 | 0 | 0 | 0
  Hypernatremia: Not Reported | 1 | 0 | 26
  Hyponatremia: Grade 0 | 24 | 29 | 5
  Hyponatremia: Grade 1 | 12 | 7 | 1
  Hyponatremia: Grade 2 | 0 | 0 | 0
  Hyponatremia: Grade 3 | 0 | 1 | 0
  Hyponatremia: Grade 4 | 0 | 0 | 0
  Hyponatremia: Not Reported | 1 | 0 | 26
  Hyperkalemia: Grade 0 | 24 | 25 | 6
  Hyperkalemia: Grade 1 | 7 | 9 | 0
  Hyperkalemia: Grade 2 | 4 | 3 | 0
  Hyperkalemia: Grade 3 | 1 | 0 | 0
  Hyperkalemia: Grade 4 | 0 | 0 | 0
  Hyperkalemia: Not Reported | 1 | 0 | 26
  Hypokalemia: Grade 0 | 24 | 25 | 6
  Hypokalemia: Grade 1 | 7 | 9 | 0
  Hypokalemia: Grade 2 | 4 | 3 | 0
  Hypokalemia: Grade 3 | 1 | 0 | 0
  Hypokalemia: Grade 4 | 0 | 0 | 0
  Hypokalemia: Not Reported | 1 | 0 | 26
  Hypercalcemia: Grade 0 | 33 | 34 | 4
  Hypercalcemia: Grade 1 | 3 | 3 | 0
  Hypercalcemia: Grade 2 | 0 | 0 | 0
  Hypercalcemia: Grade 3 | 0 | 0 | 0
  Hypercalcemia: Grade 4 | 0 | 0 | 0
  Hypercalcemia: Not Reported | 1 | 0 | 28
  Hypocalcemia: Grade 0 | 29 | 28 | 0
  Hypocalcemia: Grade 1 | 6 | 7 | 3
  Hypocalcemia: Grade 2 | 1 | 1 | 1
  Hypocalcemia: Grade 3 | 0 | 1 | 0
  Hypocalcemia: Grade 4 | 0 | 0 | 0
  Hypocalcemia: Not Reported | 1 | 0 | 28

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their randomization to study completion, (up to approximately 40 months). Serious adverse events (SAEs) and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 20 months).
Description: The number at risk for All-Cause Mortality represents all randomized participants. The number at risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Arm A: Nivolumab + Bempegaldesleukin | Arm B: Nivolumab | Arm C: Standard of Care
All-Cause Mortality (participants affected / at risk) | 8/37 | 6/37 | 12/40
Serious Adverse Events (participants affected / at risk) | 16/37 | 22/37 | 15/32
Other Adverse Events (participants affected / at risk) | 32/37 | 29/37 | 18/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivolumab + Bempegaldesleukin (N=37) | Arm B: Nivolumab (N=37) | Arm C: Standard of Care (N=32)
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 3 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0
Endocarditis noninfective (Cardiac disorders) | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0
Vallecular cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Hernial eventration (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal barrier dysfunction (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 3 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 3 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 2 | 1 | 4
Septic shock (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 1 | 3
Urosepsis (Infections and infestations) | 0 | 1 | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incision site impaired healing (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatine increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Device occlusion (Product Issues) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 3 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Immune-mediated nephritis (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivolumab + Bempegaldesleukin (N=37) | Arm B: Nivolumab (N=37) | Arm C: Standard of Care (N=32)
Anaemia (Blood and lymphatic system disorders) | 4 | 7 | 2
Eosinophilia (Blood and lymphatic system disorders) | 2 | 0 | 0
Hyperleukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 2 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 1 | 0
Hypothyroidism (Endocrine disorders) | 3 | 5 | 0
Dry eye (Eye disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 7 | 4
Diarrhoea (Gastrointestinal disorders) | 8 | 3 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 3
Oesophagitis (Gastrointestinal disorders) | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2
Asthenia (General disorders) | 9 | 5 | 1
Chills (General disorders) | 3 | 0 | 0
Fatigue (General disorders) | 8 | 6 | 3
Influenza like illness (General disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 2 | 4 | 1
Pain (General disorders) | 2 | 1 | 0
Peripheral swelling (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 10 | 3 | 4
Xerosis (General disorders) | 2 | 0 | 0
Hypersensitivity (Immune system disorders) | 3 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 2 | 1
Cystitis (Infections and infestations) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 5 | 7 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2 | 0
Amylase increased (Investigations) | 2 | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 2 | 0
Blood creatinine increased (Investigations) | 5 | 4 | 2
Gamma-glutamyltransferase increased (Investigations) | 3 | 1 | 0
Lipase increased (Investigations) | 1 | 4 | 0
Weight decreased (Investigations) | 4 | 7 | 2
Weight increased (Investigations) | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0
Headache (Nervous system disorders) | 3 | 2 | 0
Device occlusion (Product Issues) | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 2
Dysuria (Renal and urinary disorders) | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 2 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 6 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 4 | 0
Hypertension (Vascular disorders) | 1 | 6 | 0
Hypotension (Vascular disorders) | 3 | 4 | 2

LIMITATIONS AND CAVEATS:
BMS and Nektar Therapeutics jointly decided to terminate the clinical development program for bempegaldesleukin (NKTR-214) in combination with nivolumab. Discontinued survival follow-up and the stopping of submission of local labs to vendors, imaging to the BICR vendor, and PROs have resulted in confounded and incomplete trial results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT04209114/Prot_SAP_000.pdf